CLINICAL TRIAL: NCT06058650
Title: Pilot Clinical Study to Evaluate Molecular Breast Imaging- Guidance for Sampling of Breast Abnormalities
Brief Title: Molecular Breast Imaging Guidance for Breast Biopsy for Patients With Breast Abnormalities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-011329; NCI-2023-06047 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 18-011329 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2023-09-13; First posted 2023-09-28 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Breast Neoplasm
MeSH Terms: conditions — Breast Neoplasms | interventions — Technetium Tc 99m Sestamibi

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Part I (technetium Tc-99m sestamibi, MBI) (Experimental): Patients receive technetium Tc-99m sestamibi IV and undergo MBI on study.
  Interventions: Radiation: Scintimammography; Other: Technetium Tc-99m Sestamibi
- Part II (technetium Tc-99m sestamibi, MBI, biopsy) (Experimental): Patients receive technetium Tc-99m sestamibi IV and undergo MBI. Patients whose breast lesions of interest are visualized on MBI then undergo breast biopsy using the Stereo Navigator accessory.
  Interventions: Procedure: Biopsy of Breast; Other: Medical Device Usage and Evaluation; Radiation: Scintimammography; Other: Technetium Tc-99m Sestamibi

INTERVENTIONS:
Procedure: Biopsy of Breast — Undergo biopsy of breast
  Other Names: Breast Biopsy
  Arms: Part II (technetium Tc-99m sestamibi, MBI, biopsy)
Other: Medical Device Usage and Evaluation — Utilization of the Stereo Navigator accessory
  Arms: Part II (technetium Tc-99m sestamibi, MBI, biopsy)
Radiation: Scintimammography — Undergo MBI
  Other Names: Breast-Specific Gamma Imaging; MBI; Miraluma Scan; Miraluma Test; Molecular Breast Imaging; Nuclear Medicine Breast Imaging; sestamibi breast imaging; Sestamibi Scintimammography
Other: Technetium Tc-99m Sestamibi — Given IV
  Other Names: Cardiolite; Miraluma; Tc 99m Sestamibi; Tc-99m MIBI; Tc99m Sestamibi; Technetium (99mTc) Sestamibi; 99m Tc-methoxy isobutyl isonitrile

SUMMARY:
This clinical trial tests how well molecular breast imaging (MBI) works to guide the collection of a breast biopsy in patients with a breast abnormality. Currently, a biopsy is often guided by either ultrasound or mammography in order to ensure that a sample of the correct part of the breast is taken. Sometimes a lesion or part of the lesion cannot be seen on ultrasound or mammography, and, therefore, a biopsy guided with ultrasound or mammography may not be always be accurate. Studies have shown that high resolution MBI may have potential to improve the detection of some breast tumors. This trial uses a new high-resolution MBI system that may help perform a biopsy using MBI.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate a methodology for MBI-guided biopsy of suspicious breast lesions.

OUTLINE: Patients are assigned to 1 of 2 study parts.

PART I: Patients receive technetium Tc-99m sestamibi intravenously (IV) and undergo MBI on study.

PART II: Patients receive technetium Tc-99m sestamibi IV and undergo MBI. Patients whose breast lesions of interest are visualized on MBI then undergo breast biopsy using the Stereo Navigator accessory.

After completion of study intervention, patients may be asked to follow up at 3-6 months.

ELIGIBILITY:
Inclusion Criteria:

* PART I: Women aged 18 years or older
* PART I: If able to become pregnant, negative pregnancy test within 48 hours prior to MBI biopsy procedure
* PART I: Individuals who have previously (within the last 3 years) undergo an MBI study and were found to have at least one breast imaging finding on MBI that was subsequently shown (through additional imaging, biopsy or follow-up) to be benign in nature
* PART I: Individuals who have agreed to participate in the study and who have signed the study-specific informed consent
* PART II: Women aged 18 years or older
* PART II: If able to become pregnant, negative pregnancy test within 48 hours prior to MBI biopsy procedure
* PART II: Individuals who have previously (within the last 3 years) undergone an MBI study and were found to have at least one breast imaging finding on MBI that was subsequently shown (through additional imaging, biopsy or follow-up) to be benign or probably benign in nature
* PART II: Individuals who had recent conventional imaging work-up including either x-ray mammography, ultrasound, MBI, or MRI of the breast and are found to have at least one breast imaging finding for which biopsy is required or recommended, specifically:

  * Individuals who have a breast abnormality(ies) on imaging with mammography, ultrasound, MBI, or MRI (as per American College of Radiology [ACR] Breast Imaging Reporting and Data System [BIRADS] 3, or higher) and requiring imaging follow-up or biopsy confirmation
* PART II: Individuals who have agreed to participate in the study and who have signed study-specific informed consent

Exclusion Criteria:

* PART I: Women who are pregnant
* PART I: Women who are currently lactating or discontinued breastfeeding < 2 months prior to the study
* PART I: Age less than 18 years
* PART I: Women with breast implant(s) in the breast containing the lesion of interest
* PART I: Inability to provide informed consent
* PART II: Women who are pregnant
* PART II: Women who are currently lactating or discontinued breastfeeding < 2 months prior to the study
* PART II: Age less than 18 years
* PART II: Women with breast implant(s) in the breast containing the lesion of interest
* PART II: Women who have recently (within the last 3 months) undergone biopsy of the breast finding
* PART II: Women who are scheduled for a sentinel node procedure using radioactive Tc-99m within 24 hours of MBI-guided biopsy
* PART II: Patients with contraindications for core biopsy and other invasive procedures such as blood coagulation disorders, infection, or who are unwilling to discontinue use of anticoagulant medication prior to the procedure
* PART II: Inability to provide informed consent
* PART II: Women who have had surgery on the study breast(s) within the past 12 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-08-26 (Actual); Primary Completion 2026-08-26 (Estimated); Study Completion 2026-08-26 (Estimated)

PRIMARY OUTCOMES:
Validation of timeframe | Baseline
  Time from injection of the technetium Tc-99m sestamibi to identification of the appropriate needle guide hole will be reviewed to determine if and where any improvements in workflow can be made to reduce the overall procedure time for patients.
Change in image of lesion | Baseline; Up to 6 months
  The coordinates of the lesion of interest on the high resolution MBI image will be recorded. The guidance procedure will be considered successful if 1) the pre and post images of the lesion demonstrated one of the following: decreased in size, central or eccentric defect where sampled, or decrease in intensity, or 2) pathology results demonstrate malignancy or a specific benign concordant result.
Accuracy of depth estimation by difference in attenuation from opposing views | Baseline; Up to 6 months
  For each patient in whom pathology confirms successful sampling of the lesion seen on high-resolution molecular breast imaging (MBI), the error in depth estimation will be calculated as the average error for each depth estimation method from all core biopsy samples. This will allow comparison of the accuracy of the 3 different depth estimation methods and potentially provide further information on the strengths and weakness of each of the three methods for depth estimation. Uniformity activity along the entire 20 mm core would indicate failure to biopsy the lesion. Any portion of increased uptake will be noted and the center of activity will be determined relative to the mid-point of the core sample. This distance will be recorded as the difference between estimated depth and true depth.
Accuracy of depth estimation by difference in apparent lesion size | Baseline; Up to 6 months
  For each patient in whom pathology confirms successful sampling of the lesion seen on MBI, the error in depth estimation will be calculated as the average error for each depth estimation method from all core biopsy samples. This will allow comparison of the accuracy of the 3 different depth estimation methods and potentially provide further information on the strengths and weakness of each of the three methods for depth estimation. Uniformity activity along the entire 20 mm core would indicate failure to biopsy the lesion. Any portion of increased uptake will be noted and the center of activity will be determined relative to the mid-point of the core sample. This distance will be recorded as the difference between estimated depth and true depth.
Accuracy of depth estimation by triangulation | Baseline; Up to 6 months
  For each patient in whom pathology confirms successful sampling of the lesion seen on MBI, the error in depth estimation will be calculated as the average error for each depth estimation method from all core biopsy samples. This will allow comparison of the accuracy of the 3 different depth estimation methods and potentially provide further information on the strengths and weakness of each of the three methods for depth estimation. Uniformity activity along the entire 20 mm core would indicate failure to biopsy the lesion. Any portion of increased uptake will be noted and the center of activity will be determined relative to the mid-point of the core sample. This distance will be recorded as the difference between estimated depth and true depth.

CONTACTS AND LOCATIONS:
Overall Officials: Katie N. Hunt, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Hunt KN, Conners AL, Gray L, Hruska CB, O'Connor MK. Molecular Breast Imaging Biopsy with a Dual-Detector System. Radiol Imaging Cancer. 2024 Jun;6(4):e230186. doi: 10.1148/rycan.230186. PMID 38847615
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials